CLINICAL TRIAL: NCT01262612
Title: A Phase II Study of Cediranib as Palliative Treatment in Patients With Symptomatic Malignant Ascites or Pleural Effusion
Brief Title: Cediranib as Palliative Treatment in Patients With Symptomatic Malignant Ascites or Pleural Effusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO201001
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Malignant Ascites; Malignant Pleural Effusion
Keywords: cediranib; malignant ascites; malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate treatment with cediranib (Active Comparator): 8 patients with ascites and 8 patients with pleural effusion will start immediate treatment with cediranib
  Interventions: Drug: immediate cediranib
- start cediranib after 28 days BSC (Active Comparator): patients in group B will start with cediranib after one month best supportive care.
  Interventions: Drug: Start cediranib after 28 days Best Supportive Care

INTERVENTIONS:
Drug: immediate cediranib — cediranib 30 mg on day one; Special in this study is the possibility to decrease (to a minimum of 15 mg) or increase the dose (to a maximum of 30 mg oid) during the study to get an individualized optimal palliative treatment with cediranib. The patient will continue cediranib as long as a clinical benefit is experienced, independent of tumour evaluation. Each dose changes should be documented with clear reasoning and documentation of the approach taken
  Other Names: AZD2171
  Arms: immediate treatment with cediranib
Drug: Start cediranib after 28 days Best Supportive Care — patients in this group will start with cediranib after one month best supportive care. Special in this study is the possibility to decrease (to a minimum of 15 mg) or increase the dose (to a maximum of 30 mg oid) during the study to get an individualized optimal palliative treatment with cediranib. The patient will continue cediranib as long as a clinical benefit is experienced, independent of tumour evaluation. Each dose changes should be documented with clear reasoning and documentation of the approach taken.
  Other Names: AZD2171
  Arms: start cediranib after 28 days BSC

SUMMARY:
In some patients with cancer there are also cancer cells in the abdominal cavity or between the lung membranes. These cancer cells create too much moisture in the abdominal cavity or between the lung membranes. If there is fluid in the abdominal cavity (ascites fluid) this can bring on abdominal distension, abdominal pain, loss of appetite, fatigue, bloating and sometimes wheezing. Too much fluid between the lung membranes (we call this pleural fluid) gives breathlessness, chest pain and coughing. The use of diuretics may offer a small group of patients symptom reduction. Additionally, the fluid can be drained through a needle puncture or fluid collection (through a biopsy). But usually, the moisture quickly returns.

Previous research done in this hospital with cediranib showed that with some patients with cancer who suffered from fluid in the abdominal cavity or between the lung membranes, this moisture reduces while using this drug. It also reduced the symptoms caused by this excessive moisture.

The current study is conducted to see whether patients with cancer and fluid in the abdominal cavity or fluid between the lung blades benefit from using cediranib. This involves not only whether the amount moisture reduces, but also if the complains decrease. In addition, we will carefully consider the possible side effects of cediranib.

DETAILED DESCRIPTION:
Malignant ascites is a difficult clinical problem. Increasing intra-abdominal pressure resulting from fluid accumulation may cause anorexia, sleep disturbance, pain, dyspnoea, abdominal distension, fatigue, nausea vomiting and reduced mobility. The main complaints of pleural effusion are dyspnoea and cough. Paracentesis and thoracentesis provide relief for a very limited period.

Studies have shown high concentrations of VEGF in malignant ascites and pleural effusion. Beneficial effects of treatment with an intravenous or intraperitoneal antibody against VEGF on malignant ascites have been reported. In the recent past we have treated two patients with symptomatic malignant ascites (colorectal cancer and ovarian cancer, respectively) in a phase I study with cediranib. Shortly after start of cediranib, within a couple of days, the ascites disappeared. However, after stopping cediranib for progressive disease on other sites the ascites reappeared within days. Therefore, one of those patients was treated with cediranib as palliative treatment until two days before his death, which was beneficial for this patient.

In this phase II study we would like to investigate the effects of treatment with cediranib as palliative treatment on malignant ascites or pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic malignant ascites and/or pleural effusion (from a histological proven solid malignancy which is refractory to standard anti-tumour therapy of for which no standard therapy exists)
* Karnofsky score ≥ 50 if the low performance score is due to ascites and/or pleural effusion, otherwise ≥ 60
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

Contraindications for treatment with cediranib:

* The presence of a pleural or peritoneal tap
* Untreated unstable brain or meningeal metastases.
* Previous treatment with chemotherapeutic agents or tyrosine kinase inhibitors (TKIs) within 14 days prior to the first dose of cediranib, with cetuximab within 30 days prior to the first dose of cediranib, or with bevacizumab within 60 days prior to the first dose of cediranib
* Inadequate bone marrow reserve as demonstrated by an absolute neutrophil count ≤1.5 x 109/L or platelet count ≤100 x 109/L
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2,5 x ULN
* Serum creatinine > 1.5 x ULRR or a creatinine clearance of ≤ 50mL/min calculated by Cockcroft-Gault
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart unless urinary protein < 1.5g in a 24 hr period
* Prothrombin time (PT) and activated partial thromboplastin time (APTT) > 2 x ULN History of significant gastrointestinal impairment, as judged by the Investigator, that would significantly affect the absorption of cediranib, including the ability to swallow the tablet whole. Patients with an ileostoma.
* Patients with a history of poorly controlled hypertension with resting blood pressure >150/100 in the presence or absence of a stable regimen of anti-hypertensive therapy. Patients who are currently receiving maximal doses of calcium channel blockers or more than 1 antihypertensive for the treatment of hypertension are also ineligible.
* Any evidence of severe or uncontrolled diseases e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease.
* Unresolved toxicity > CTC grade 1 from previous anti-cancer therapy (including radiotherapy) except alopecia (if applicable) or polyneuropathy.
* Mean QTc with Bazetts correction >470msec in screening ECG or history of familial long QT syndrome
* Significant haemorrhage (>30mL bleeding/episode in previous 3 months) or haemoptysis (>5mL fresh blood in previous 4 weeks)
* Recent (<14 days) major surgery prior to entry into the study, or a surgical incision that is not fully healed
* Pregnant or breast-feeding women or women of childbearing potential with a positive pregnancy test prior to receiving study medication
* Known risk of the patient transmitting HIV, hepatitis B or C via infected blood
* Treatment with an investigational (non-registered) drug within 30 days prior to the first dose of cediranib
* Other concomitant anti-cancer therapy (including LHRH agonists) except steroids
* Concomitant use of any medication that may significantly affect hepatic cytochrome P450 drug metabolising activity by way of enzyme induction (e.g., phenytoin) or inhibition (e.g., ketoconazole, ritonavir, erythromycin) within 2 weeks if the first dose of cediranib and throughout the study period
* Patients being treated with anticoagulants (with the exception of low molecular weight heparin).
* Patients previously treated with anthracyclines (total of > 550 mg/m2 doxorubicine) and an ejection fraction on the MUGA scan below 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
puncture free survival | 44 days
  If the puncture free survival after start of treatment with cediranib (time to first need for paracentesis or thoracentesis or time to death, which event occurred first) is more than 44 days the treatment of ascites and/or pleural effusion with cediranib is effective.

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, Md PhD, Principal Investigator — University Medical Centre Nijmegen
Locations (1):
- University Medical Centre Nijmegen, Nijmegen, Gelderland, Netherlands